CLINICAL TRIAL: NCT04769843
Title: Incorporating the Psychological Consequences of Dysphagia Into Swallowing Care: A Preliminary Investigation
Brief Title: Impact of Swallowing Impairment on Individuals With Parkinson Disease
Status: Completed | Type: Observational
Sponsor: Northern Arizona University (Other)
Responsible Party: Principal Investigator, Rebecca Bartlett, Assistant Professor, Northern Arizona University
Other Study IDs: 1508794
Record Dates: First submitted 2021-02-19; First posted 2021-02-25 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease; Dysphagia
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this online study, investigators will explore the psychosocial burdens of swallowing difficulties in people with Parkinson's Disease. This study is completely virtual, so you can participate from wherever you live in the United States. Participation requires you to complete a one-hour Zoom interview and a brief questionnaire. You will be compensated with a $25 Walmart gift card. To learn more, please use the "send email" feature. Thank you!

DETAILED DESCRIPTION:
This is a mixed methods study. The investigators will collect qualitative data from participants by conducting 1-2 hour semi-structured interviews on Zoom. The interview questions are designed to systemically inquire about patient experiences, affective reactions, coping strategies, social support, self-identity issues, and treatment experiences. The investigators will collect quantitative data by asking participants to complete The Brief Illness Perception Questionnaire. The data will be analyzed using a comprehensive stress and coping model, which has not been done previously in the field. The investigators hope to discover themes about psychosocial burdens and related coping mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Participants must currently have oropharyngeal dysphagia and Parkinson Disease
* Participants must be at least 18 years of age
* Participants must speak English.

Exclusion Criteria:

* Participants whose receptive and expressive language skills will not allow them to participate in one-on-one interviews

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from 1) local Parkinson Disease support groups, 2) through referrals from local speech-language pathologists, and 3) through the Fox Trial Finder on the Michael J. Fox Foundation website.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of the Impact of Swallowing Impairment on Individuals with Parkinson Disease as Expressed During Interviews | To be assessed from the participant interviews through study completion, an average of 1 year.
  A 1-2 hour, semi-structured interview will be conducted with each participant on Zoom to identify patient experiences, affective reactions, coping strategies, social support, self-identity issues, and treatment experiences associated with swallowing impairment.

SECONDARY OUTCOMES:
Overall Score on Brief Illness Perception Questionnaire (Brief IPQ) as Self-Reported by Participants | The Brief IPQ will be mailed to participants after their interview and asked to complete it and return it to us within one week.
  The Brief IPQ is a self-report survey that contains nine items that quantify the cognitive and emotional representations of an illness. It has good test-retest reliability and concurrent validity with relevant measures in a few populations with chronic disease. Scores range from 0 (i.e., illness has no effect on life) to 80 points (i.e., illness extremely effects various aspects of life).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca S Bartlett, PhD, Principal Investigator — Northern Arizona University
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT04769843/ICF_000.pdf